CLINICAL TRIAL: NCT04310046
Title: Optimal Timing of Transcatheter Aortic Valve Implantation and Percutaneous Coronary Intervention - The TAVI PCI Trial
Acronym: TAVI-PCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAVI PCI
Record Dates: First submitted 2020-02-12; First posted 2020-03-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Aortic Stenosis; Coronary Artery Disease; TAVI; PCI
Keywords: Aortic Stenosis; Transcatheter Aortic Valve Replacement; Percutaneous Coronary Intervention; Heart Diseases; Valvular Disease; Coronary Artery Disease; Myocardial Ischemia; Cardiovascular Diseases; Vascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease; Heart Diseases; Myocardial Ischemia; Cardiovascular Diseases; Vascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCI before TAVI (Other): PCI is performed within 1-45 days before TAVI.
  Interventions: Procedure: PCI before TAVI
- PCI after TAVI (Experimental): PCI is performed within 1-45 days after TAVI.
  Interventions: Procedure: PCI after TAVI

INTERVENTIONS:
Procedure: PCI before TAVI — TAVI is performed using the Edwards SAPIEN Transcatheter Heart Valve®. PCI is performed in any suitable lesion with ≥70% diameter stenosis on coronary angiography in a coronary artery ≥2.5 mm in diameter.
  Arms: PCI before TAVI
Procedure: PCI after TAVI — TAVI is performed using the Edwards SAPIEN Transcatheter Heart Valve®. PCI is performed in any suitable lesion with ≥70% diameter stenosis on coronary angiography in a coronary artery ≥2.5 mm in diameter.
  Arms: PCI after TAVI

SUMMARY:
The primary objective of this study is to compare, in patients with severe aortic stenosis and concomitant coronary artery disease accepted for transcatheter aortic valve implantation (TAVI) and percutaneous coronary intervention (PCI) by the multidisciplinary Heart Team, the safety and efficacy of angiography-guided complete revascularization performed after (within 1-45 days) with angiography-guided complete revascularization performed before (within 1-45 days) TAVI using the Edwards SAPIEN Transcatheter Heart Valve®.

DETAILED DESCRIPTION:
The prevalence of coronary artery disease in patients with severe aortic stenosis is high. About 30-60% of patients undergoing TAVI exhibit coexisting coronary artery disease. Optimal timing of coronary revascularization in patients with severe aortic stenosis and concomitant coronary artery disease undergoing TAVI is uncertain.

The goal of this investigator-initiated, randomized, multicenter, two-arm, open-label, non-inferiority trial is to compare two treatment strategies that are currently performed in clinical practice: PCI before TAVI versus PCI after TAVI in patients with severe aortic stenosis and concomitant coronary artery disease.

In this trial, patients with severe aortic stenosis and concomitant coronary artery disease accepted for TAVI and PCI by the Heart Team will be randomized in a 1:1 ratio to the following strategies: angiography-guided complete coronary revascularization before (within 1-45 days) or after (within 1-45 days) TAVI using the Edwards SAPIEN Transcatheter Heart Valve®.

For both treatment groups, coronary artery lesions with ≥70% diameter stenosis on coronary angiogram (by visual estimation) in a coronary artery ≥2.5 mm in diameter are considered significant.

TAVI and PCI will be performed according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years with severe aortic stenosis and concomitant coronary artery disease accepted for transfemoral TAVI with an Edwards SAPIEN Transcatheter Heart Valve™ and PCI by a multidisciplinary Heart Team.
2. Severe aortic stenosis defined as aortic valve area (AVA) ≤1.0 cm2 and/or mean pressure gradient ≥40 mmHg (echocardiography) and at least one of the following criteria:

   1. Dyspnea
   2. Angina symptoms
   3. Syncope
   4. Decline in left ventricular ejection fraction <50%, symptoms or fall in blood pressure on exercise testing, or presence of high-risk criteria (peak transaortic velocity >5.5 m/s, severe valve calcification, peak transaortic velocity progression ≥0.3 m/s per year, or severe pulmonary hypertension with systolic pulmonary artery pressure >60 mmHg) according to current guidelines.
3. At least one coronary artery lesion with ≥70% diameter stenosis on coronary angiogram (by visual estimation) in a coronary artery ≥2.5 mm in diameter and Thrombolysis in Myocardial Infarction (TIMI) flow grade III, deemed amenable to PCI within 45 days before or after TAVI. Hemodynamic lesion assessment by fractional flow reserve (FFR), instantaneous wave-free ratio (iwFR), or comparable indices as well as intravascular imaging-guided PCI are left at the discretion of the operator.
4. Written informed consent.

Exclusion Criteria:

1. TAVI by transapical, subclavian, or transaortic access
2. Admission with acute myocardial infarction within 30 days before randomization
3. Elective coronary revascularization within 3 months before randomization
4. Previous coronary artery bypass grafting (CABG)
5. Syntax Score I ≥33
6. Any contraindications for dual antiplatelet therapy with aspirin and a P2Y12 inhibitor (clopidogrel, ticagrelor or prasugrel), except for patients on oral anticoagulation
7. Planned open heart surgery
8. Known pregnancy at the time of inclusion
9. Life expectancy <1 year due to other severe non-cardiac disease
10. Participation in another clinical study with an investigational product
11. Acute COVID-19 infection
12. Patient with previously treated aortic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the number of participants experiencing the primary outcome measure | 1 year
  The primary outcome measure is a composite of:
  * All-cause death
  * Non-fatal myocardial infarction
  * Ischemia-driven revascularization
  * Rehospitalization (valve- or procedure-related including heart failure)
  * Life-threatening/disabling or major bleeding (according to VARC-2)

SECONDARY OUTCOMES:
The primary outcome measure | Discharge (hospitalization first and second procedure), 3 months, 2 years and 5 years
Single components of the primary endpoint | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
All cause death and myocardial infarction | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Cardiovascular death and myocardial infarction | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
All cause death, myocardial infarction and ischemia-driven revascularization | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
All cause death, myocardial infarction, ischemia-driven revascularization and rehospitalization | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Cardiovascular death | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Stroke | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Peri-procedural myocardial infarction (PCI) | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Peri-procedural myocardial infarction (TAVI) | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Major vascular complications | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Bleeding events | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
  Bleeding events are defined according to the Bleeding Academic Research Consortium (BARC) definition
Symptom status and change from baseline in symptom status (Canadian Cardiovascular Society (CCS) and New York Hear Association (NYHA) classification) | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Quality of life (as assessed by the KCCQ and TASQ questionnaires) | Admission (for second procedure), 3 months, 1 year, 2 years and 5 years
  Kansas City Cardiomyopathy questionnaire (KCCQ) and the Toronto Aortic Stenosis Quality of Life questionnaire (TASQ)
Change from baseline in Quality of life (as assessed by the KCCQ and TASQ questionnaires) | Admission (for second procedure), 3 months, 1 year, 2 years and 5 years
  Kansas City Cardiomyopathy questionnaire (KCCQ) and the Toronto Aortic Stenosis Quality of Life questionnaire (TASQ)

OTHER OUTCOMES:
Procedural success (PCI) | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Device success (TAVI) | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Any revascularization | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Target lesion revascularization | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Target vessel revascularization | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
In-stent thrombosis | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Acute kidney injury | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
New-onset atrial fibrillation | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
New permanent pacemaker implantation | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Aortic valve-related dysfunction requiring repeat procedure | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Amount of contrast medium (PCI) | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Fluoroscopy time (PCI) | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Radiation exposure (dose area product, PCI) | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Conversion to open heart surgery | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years
Use of catecholamines during PCI | Discharge (hospitalization first and second procedure), 3 months, 1 year, 2 years and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Markus Kasel, MD, Principal Investigator — University Hospital, Zürich; Barbara E. Stähli, MD, eMBA, Principal Investigator — University Hospital, Zürich
Locations (1):
- University Hospital Zürich, Cardiology Department, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No